CLINICAL TRIAL: NCT02672488
Title: Safety and Efficacy of Metformin Plus Sorafenib as First-line Therapy in Patients With Advanced Hepatocellular Carcinoma(BCLC-C): A Phase 2 Randomized Study
Brief Title: Metformin Plus Sorafenib for Advanced HCC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: First Affiliated Hospital of Harbin Medical University (Other); Harbin Medical University (Other); Liaoning Cancer Hospital & Institute (Other); Shanghai Zhongshan Hospital (Other); Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: METSOR
Record Dates: First submitted 2015-12-07; First posted 2016-02-03 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2015-12

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sorafenib and Metformin (Experimental): Sorafenib 400μg tablet by mouth and Metformin 500mg tablet by mouth with meal, twice per day
  Interventions: Drug: Sorafenib; Drug: Metformin
- Sorafenib Alone (Active Comparator): Sorafenib 400μg tablet by mouth, twice per day
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Sorafenib — Standard treatment for advanced HCC
  Other Names: Nexavar
Drug: Metformin — To evaluate the safety and efficacy of the combined treatment of Metformin and Sorafenib for advanced HCC
  Other Names: Glucophage
  Arms: Sorafenib and Metformin

SUMMARY:
Metformin is a widely used oral drug for type 2 diabetes and its antitumor effects have got much more attentions recently. It has been shown that metformin exerts anti-cancer activities in several cancers, including primary liver cancer. In this phase II study, safety and efficacy of the combination of metformin and sorafenib will be evaluated in patients with advanced hepatocellular carcinoma.

DETAILED DESCRIPTION:
Sorafenib is the standard choice for advanced hepatocellular carcinoma (BCLC-C), but the efficacy is not satisfied. Metformin is a widely used oral drug for type 2 diabetes and its antitumor effects have got much more attentions recently. It has been shown that metformin exerts anti-cancer activities in several cancers, including primary liver cancer. Recent studies suggest that metformin treatment can reduce the risk of HCC in patients with type 2 diabetes and inhibit HCC invasion and increase drug sensitivity to sorafenib, however, the safety and efficacy of combined therapy for advanced hepatocellular carcinoma remains unclear. In this phase II study, patients with advanced hepatocellular carcinoma, measurable disease, and an Eastern Cooperative Oncology Group performance score≤1 will be enrolled. Eligible subjects will be randomly assigned to receive the treatment of sorafenib or metformin plus sorafenib. The potential improvement of overall survival, time to progression and safety will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Ability of the research subject or authorized legal representative to understand and the willingness to sign a written informed consent document
2. Confirmed hepatocellular carcinoma according to one of following three criteria:

   histopathology,Two radiographic techniques (US, MRI, CT, or Angiography) that confirm lesion with typical arterial hypervascularization,Barcelona Clinical Liver Cancer staging C (BCLC-C)
3. Age > 18 years old
4. Patients with liver disease classified as Child Pugh class A
5. Eastern Clinical Oncology Group (ECOG) performance status 0，1 or 2 (Appendix I)
6. Hemoglobin ≥ 9 g/dL
7. Absolute Neutrophil count（ANC）≥ 1,500 /mm3
8. Platelet count≥ 50,000 /ul
9. Total Bilirubin < 2 mg/dL
10. Transaminases (SGOT and SGPT) no more than 5 times the upper limit of normal
11. Alkaline phosphatase < 4 times the upper limit of normal
12. Both men and women and members of all races and ethnic groups are eligible for this study
13. Prothrombin time > 50% 或 PT-INR < 2.3

Exclusion Criteria:

1. Child Pugh Score is 7 with ascites
2. Severe cardiovascular disease
3. Uncontrollable hypertension
4. History of HIV infection
5. Active clinical severe infection（>grade 2 ，NCI-CTCAE Version3.0）
6. Women who are pregnant
7. Administration of any systemic chemotherapy within the last 6 months
8. Presence of History of gastrointestinal bleeding before randomization
9. Epileptic seizures requiring drug therapy
10. History of allograft transplantation
11. Patients with signs of bleeding or medical history
12. Patients undergoing kidney dialysis
13. Metastatic liver cancer
14. Uncontrollable ascites
15. Encephalopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 12 months or time to death

SECONDARY OUTCOMES:
Time To Progression | 12 months or time to death
Progression Free Survival | 12 months
Objective Response Rate | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ti Zhang, MD, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: Yes